CLINICAL TRIAL: NCT05632133
Title: a Randomized Pilot Study of Lacosamide's Effect on Calcitonin Gene-related Peptide in Migraine Patients
Brief Title: The Lacosamide's Effect on Calcitonin Gene-related Peptide in Migraine Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, prinicipal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2398816
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Effect of Drug; Migraine Disorders
Keywords: migraine; lacosamide; Egypt
MeSH Terms: conditions — Migraine Disorders | interventions — Lacosamide; Tablets; Ibuprofen

STUDY DESIGN:
Intervention Model Description: We assessed CGRP before and after treatment in two groups of episodic migraine patients; the first group (the lacosamide group) received Ibuprofen 200-400 mg as a treatment for acute migraine attacks and 50 mg lacosamide Bid for 3 months, and the second group (control group) received only Ibuprofen 200-400 mg as a treatment for acute migraine attacks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lacosamide group (Experimental): We assessed the serum level of CGRP before and after 3 months of treatment in 100 episodic migraine patients receiving 50 mg lacosamide Bid and Ibuprofen 200-400 mg only during migraine attacks.
  Interventions: Drug: Lacosamide 50 MG Oral Tablet; Drug: Ibuprofen 400 mg
- control group (Experimental): We assessed the serum level of CGRP before and after 3 months of treatment in 100 episodic migraine patients receiving Ibuprofen 200-400 mg only during migraine attacks.
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Lacosamide 50 MG Oral Tablet — We assessed the serum level of CGRP before and after 3 months of treatment in 100 episodic migraine patients receiving 50 mg lacosamide Bid and Ibuprofen 200-400 mg only during migraine attacks.
  Arms: lacosamide group
Drug: Ibuprofen 400 mg — We assessed the serum level of CGRP before and after 3 months of treatment in 100 episodic migraine patients receiving Ibuprofen 200-400 mg only during migraine attacks.
  Other Names: control

SUMMARY:
We assessed serum CGRP concentrations before and after treatment in two hundred episodic migraine patients according to the International Classification of Headache Disorders 3rd edition, aged 10-55 years. We divided them into two groups first one received Ibuprofen 200-400 mg as a treatment for acute migraine attacks and lacosamide 50 mg Bid for 3 months, and the other group received only Ibuprofen 200-400 mg as a treatment for acute migraine attacks.

DETAILED DESCRIPTION:
Two hundred episodic migraine patients, according to the International Classification of Headache Disorders 3rd edition, aged 10-55 years with migraines. We divided them into two groups first one received Ibuprofen 200-400 mg as a treatment for acute migraine attacks and lacosamide 50 mg Bid for 3 months, and the other group received only Ibuprofen 200-400 mg as a treatment for acute migraine attacks. Our selected patients were naive and didn't receive any other prophylactic therapy for migraine.

for each patient, the investigators did

1. detailed history taking with stress on Age, sex, and criteria and type of migraine
2. general examination
3. full neurological examination: Full neurological examination
4. Laboratory investigations include: Serum creatinine, Liver functions test to exclude any metabolic disorder.
5. Approximately 5 ml of venous blood was drawn from all participants and centrifuged at 1000×g for 10 min. Serums were separated from the blood sample and stored at - 20 ℃. The serum calcitonin gene-related peptide (CGRP) concentrations will be measured by adapting the enzyme-linked immunosorbent assay (ELISA) kit following manufacturer protocols.
6. Serum level CGRP before starting treatment and after three months of treatment
7. MRI T1, T2, and flair to exclude any secondary cause of headache.

ELIGIBILITY:
Inclusion Criteria:

* Naive migraine patients according to the International Classification of Headache Disorders 3rd edition aged 10-55 years,

Exclusion Criteria:

* Patients with major neurological disorders such as ( epilepsy, ischemic or hemorrhagic stroke, multiple sclerosis, mitochondrial diseases, brain tumors, and patients with essential tremors.
* patients with major systemic diseases such as malignancy, collagen diseases, liver diseases, and renal diseases.
* patients with cardiovascular diseases like hypertension (systolic blood pressure of more than 130 and/or diastolic blood pressure of more than 85 mm/Hg on at least three different occasions, diabetes (fasting plasma glucose level >126 mg/dl and/or a casual plasma glucose >200 mg/dl and/or HbA1C more than 6.5.
* patients with valvular and ischemic heart diseases,
* patients who received prophylactic treatment for migraine,
* patients with any contraindications to lacosamide.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
serum CGRP level in lacosamide and control groups | 3 months
  Approximately 5 ml of venous blood was drawn from all participants and then centrifuged at 1000×g for 10 min. Serums were separated from the blood sample and stored at - 20℃.
  The serum CGRP concentration was measured before starting treatment and after 3 months of treatment by adapting the enzyme-linked immunosorbent assay (ELISA) kit following manufacturer protocols.

SECONDARY OUTCOMES:
efficacy of lacosamide | 3 months
  We compared the monthly migraine days change in both the lacosamide and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD,PHD, Study Director — neurology department kafr el-sheikh university; mohamed G. Zeinhom, PHD, Principal Investigator — neurology department kafr el-sheikh university; sherihan R. Ahmed, MSc, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All the data supporting this research's findings may be available from the principal investigator Mohamed G. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Result] Collins JJ, Baase CM, Sharda CE, Ozminkowski RJ, Nicholson S, Billotti GM, Turpin RS, Olson M, Berger ML. The assessment of chronic health conditions on work performance, absence, and total economic impact for employers. J Occup Environ Med. 2005 Jun;47(6):547-57. doi: 10.1097/01.jom.0000166864.58664.29. PMID 15951714
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523
- [Result] Mushet GR, Miller D, Clements B, Pait G, Gutterman DL. Impact of sumatriptan on workplace productivity, nonwork activities, and health-related quality of life among hospital employees with migraine. Headache. 1996 Mar;36(3):137-43. doi: 10.1046/j.1526-4610.1996.3603137.x. PMID 8984084
- [Result] Landy S, DeRossett SE, Rapoport A, Rothrock J, Ames MH, McDonald SA, Burch SP. Two double-blind, multicenter, randomized, placebo-controlled, single-dose studies of sumatriptan/naproxen sodium in the acute treatment of migraine: function, productivity, and satisfaction outcomes. MedGenMed. 2007 Jun 7;9(2):53. PMID 17955107
- [Derived] Elgamal S, Ahmed SR, Nahas MM, Hendawy SR, Elshafei O, Zeinhom MG. The effect of lacosamide on calcitonin gene-related peptide serum level in episodic migraine patients: a randomized, controlled trial. Acta Neurol Belg. 2024 Jun;124(3):965-972. doi: 10.1007/s13760-024-02499-9. Epub 2024 Mar 19. PMID 38502425